CLINICAL TRIAL: NCT00961597
Title: Repair of Human Meniscus Complex Red/White Tears With or Without Platelet-Rich Plasma
Brief Title: Assessment of Outcome of Meniscus Repair With or Without Platelet Rich Plasma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sue Barber-Westin (Other)
Responsible Party: Sponsor-Investigator, Sue Barber-Westin, Director Clinical Studies, Cincinnati Sportsmedicine Research and Education Foundation
Organization: Cincinnati Sportsmedicine Research and Education Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MenisPRP-001
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Cartilage Disease
Keywords: Meniscus; Avascular region; Platelet rich plasma
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meniscus repair with PRP (Experimental): Meniscus repair for tears extending into the red/white region with PRP
  Interventions: Procedure: Meniscus repair with PRP
- Meniscus repair without PRP (Active Comparator)
  Interventions: Procedure: Meniscus repair for red/white tears without PRP

INTERVENTIONS:
Procedure: Meniscus repair for red/white tears without PRP — Same operation as experimental, only without the use of platelet rich plasma.
  Arms: Meniscus repair without PRP
Procedure: Meniscus repair with PRP — Meniscus repair with platelet rich plasma using vertical divergent suture techniques.
  Arms: Meniscus repair with PRP

SUMMARY:
The purpose of this investigation is to determine the clinical outcome of repair of meniscus tears located in the "red/white" region using a well-known suture technique combined, when indicated, with platelet-rich plasma to enhance healing. The outcome of this operation will be determined in a consecutive group of patients with an established, rigorous knee rating system a minimum of 2 years postoperatively. Results will be determined by the analysis of subjective and functional factors, sports and occupational activity levels, a comprehensive physical examination, and a radiographic evaluation using standard plain x-rays and magnetic resonance imaging. The investigators hypothesize that meniscus repairs will significantly reduce tibiofemoral compartment pain and allow for increased knee function and activity levels. The platelet rich plasma adjunct will be used in complex meniscus tears in which a portion of the tear extends into the avascular region classified as either longitudinal, horizontal, or radial. The investigators hypothesize that the healing rate of these repairs will be superior to those previously reported in clinical studies in patients who had the suture repair technique alone.

DETAILED DESCRIPTION:
There are many published clinical studies of complex meniscus tears in the red/white region with success rates that vary from 57% to 100%. Meniscus repairs that fail in this region usually require subsequent removal, which essentially results in loss of the majority of meniscal function and risk of future disabling osteoarthritis. This study will determine if the addition of platelet rich plasma increases the success rate of complex meniscus repairs of longitudinal, horizontal, or radial tears in the red-white region. The investigators have over two decades of experience with clinical studies of meniscus repairs in patients whose age ranged from 9 to 58 years. Those investigations revealed an average success rate in terms of retention of meniscus tissue of 80%. However, meniscus tears classified as horizontal, radial, double longitudinal, and complex multiplanar had success rates of 71-73% which prompted the need for an adjunct therapeutic measure, such as platelet rich plasma, to increase the healing potential in these cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for meniscus repair who provide informed consent to participate

Exclusion Criteria:

* Patients scheduled for meniscus repair who refuse to participate
* Presence of a tumor, metastatic disease, active infections, platelet count < 10 5/hl Hgb < 10 g/dl, pregnancy, active breastfeeding, and allergy to Bupivicaine
* Patients with preexisting thrombocytopenia, hypofibrinogenemia, or who are on anti-coagulant therapy, or who have a potential hypersensitivity to bovine products

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Elimination of pain | Minimum 2 years postoperatively

SECONDARY OUTCOMES:
Magnetic resonance imaging: T2 mapping, signal changes | Minimum 2 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Noyes, M.D., Principal Investigator — Cincinnati Sportsmedicine Research and Education Foundation
Locations (1):
- Cincinnati Sportsmedicine and Orthopaedic Center, Cincinnati, Ohio, United States